CLINICAL TRIAL: NCT05935644
Title: ORCHID: A Novel Positive Affect Intervention for Aging, Racial/Ethnic Minoritized Women With HIV (Miami)
Brief Title: ORCHID: An Online Intervention for Persons With HIV (Miami)
Acronym: ORCHID-Miami
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Lunthita M. Duthely, Research Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20221247
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: HIV/AIDS; HPV Infection
Keywords: depression; mobile applications; cortisol levels
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Papillomavirus Infections; Depression | interventions — Benzethonium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ORCHID Group (Experimental): Participants in the ORCHID group will receive an online intervention that improves depressive symptoms and positive affect (emotions) for clinic-based persons living with HIV, for up to 6 months.
  Interventions: Behavioral: ORCHID

INTERVENTIONS:
Behavioral: ORCHID — The intervention includes 8 modules, which are delivered online, approximately 30 minutes per session, and participants will engage a minimum of once per week. Participants may also meet online or in-person with a navigator, up to 4 times.

SUMMARY:
The purpose of this research is to test ORCHID (Optimizing Resilience & Coping with HIV through Internet Delivery), a skills-building intervention that improves mental health status for persons with HIV, who are at-risk for falling out of care.

ELIGIBILITY:
Inclusion Criteria:

1. Cis-gender women,
2. Receiving human immunodeficiency virus (HIV) care at the University of Miami Women's HIV Service,
3. Recent history (12-month) of cervical or anal dysplasia or human papilloma virus (HPV) positivity; AND a recent (12-month) history of one or more of the following:

i) drug use (alcohol, tobacco products, marijuana, illicit drugs) or ii) depression or iii) psychiatric condition (anxiety, post-traumatic stress disorder (PTSD)) or iv) unsuppressed HIV viral load d. All life stages - pregnant, non-pregnant, pre/post-menopausal

Exclusion Criteria:

1. Under 18
2. Not able to read/write English at the 6th grade level
3. Cognitively impaired adults (as documented in medical records)
4. Debilitating psychiatric condition (e.g. schizophrenia/bi-polar/psychotic disorders)
5. Prisoners

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-27 (Estimated); Study Completion 2025-10-27 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants who Complete ORCHID | Up to 6 months
  Average across all participants of the proportion of participants who login to all 8 ORCHID intervention sessions, calculated as total number of sessions opened (0-8) divided by 8.

SECONDARY OUTCOMES:
Depression as measured by Patient Health Questionnaire (PHQ-9) | Up to 6 months
  Depression will be measured using the PHQ-9 (range 0 to 27), higher scores indicate higher levels of depressive symptoms
Positive Affect as measured by Positive and Negative Affect Schedule (PANAS) | Up to 6 months
  Positive affect will be measured using the PANAS, range is 10 to 50, higher scores indicate higher levels of positive emotions.

CONTACTS AND LOCATIONS:
Overall Officials: Lunthita M Duthely, Ed.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No